CLINICAL TRIAL: NCT02563795
Title: Does the Reduction of Local Anesthetic Dose Provide Surgical Anesthesia While Avoiding Maternal Hypotension in Obese Pregnant for C/S by Single Shot Spinal Anesthesia?
Brief Title: Low Dose Spinal Anesthesia in Cesarean Surgery
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, MD, Ankara University
Other Study IDs: ANK-42479
Record Dates: First submitted 2015-09-18; First posted 2015-09-30 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Maternal Hypotension; Anesthesia
Keywords: Spinal anesthesia; Cesarean; Maternal hypotension
MeSH Terms: interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group I: Pregnant with BMI<30 and having spinal anesthesia with 10 mg hyperbaric bupivacaine
  Interventions: Drug: Bupivacaine
- Group II: Pregnant with BMI<30 and having spinal anesthesia with 7,5 mg hyperbaric bupivacaine+25 mcg fentanyl
  Interventions: Drug: Fentanyl
- Group III: Pregnant with BMI>30 and having spinal anesthesia with 10 mg hyperbaric bupivacaine
  Interventions: Drug: Bupivacaine
- Group IV: Pregnant with BMI>30 and having spinal anesthesia with 7,5 mg hyperbaric bupivacaine+25 mcg fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Bupivacaine — To compare low dose spinal anesthesia with bupivacaine alone if it can maintain surgical anesthesia during cesarean section in obese and non-obese pregnants
  Other Names: Fentanyl
  Groups: Group I; Group III
Drug: Fentanyl — To compare low dose spinal anesthesia with bupivacaine+ fentanyl alone if it can maintain surgical anesthesia during cesarean section in obese and non-obese pregnants
  Other Names: Bupivacaine
  Groups: Group II; Group IV

SUMMARY:
Anesthesia for cesarean section requires special importance because it may affect both mother and the baby. To avoid maternal hypotension related to spinal anesthesia must be the primary objective during anesthesia. Even though many factors influence sensory nerve block for surgical anesthesia, local anesthetic dose is the main determinant. Another factor that influence the sensory nerve block is the obesity related to pregnancy. Due to the enlargement of epidural venous plexus related to pregnancy, the subarachnoid and epidural space reduces, so the local anesthetic requirement also reduces. Many investigators recommend lower dose of local anesthetic in obese patients due to reduced requirement There are many studies about dose regimens for cesarean anesthesia, but ideal dose have not been found. Investigators have designed this study to see the effects of conventional dose (10 mg bupivacaine) vs. low dose plus fentanyl (7,5 mg bupivacaine+25 mcg fentanyl) in obese and normal weight pregnant for cesarean section. The hypothesis was: the low dose regimen provides surgical anesthesia in obese patients while avoiding maternal hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients

Exclusion Criteria:

* Spinal anesthesia contraindications, thrombocytopenia, coagulation defects, cardiomyopathy, placenta previa, twin pregnancy, hypersensitivity to amide local anesthetics or fentanyl, infection at the injection site, neurologic disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing cesarean section under spinal anesthesia in obstetric clinic
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
VAS score < 6 with only spinal anesthesia | Approximately 30 min, during surgery
  Achieving surgical anesthesia with low dose spinal anesthesia in obese pregnants

SECONDARY OUTCOMES:
Maternal hypotension | Approximately 30 min, during surgery
  Avoiding maternal hypotension

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIM GUCLU, MD, Principal Investigator — Ankara University
Locations (1):
- Cigdem Yildirim Guclu, Ankara, Turkey (Türkiye)